CLINICAL TRIAL: NCT07177365
Title: ICBT Clinical Validation - A Clinical Study on Internet-based Cognitive Behavioral Intervention for Generalized Anxiety Disorder and Major Depressive Disorder
Brief Title: Internet-Based Cognitive Behavioral Therapy With Treatment as Usual for Generalized Anxiety Disorder and Major Depressive Disorder in Taiwan (ICBT-TW)
Acronym: ICBT-TW
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202506094RSPD; C114B0B014500 (Other Grant/Funding Number: National Health Research Institutes, Taiwan)
Record Dates: First submitted 2025-09-15; First posted 2025-09-17 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-08

CONDITIONS: Generalized Anxiety Disorder (GAD); Major Depressive Disorder (MDD)
Keywords: Internet-Based Cognitive Behavioral Therapy; ICBT; Digital Mental Health; Online Therapy; Randomized Controlled Trial; Cognitive Restructuring; Mindfulness; Self-Compassion; Taiwan; Treatment as Usual (TAU)
MeSH Terms: conditions — Generalized Anxiety Disorder; Depressive Disorder, Major | interventions — Therapeutics; Single Person

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAU + ICBT (Experimental): Participants will receive standard psychiatric care (Treatment as Usual, TAU) plus an 8-week Internet-based Cognitive Behavioral Therapy (ICBT) program delivered via the National Health Research Institutes platform.
  Interventions: Behavioral: Internet-Based Cognitive Behavioral Therapy (ICBT)
- TAU Only (Active Comparator): Participants will receive standard psychiatric care (TAU) without ICBT during the study period. After study completion, they may request access to the ICBT program.
  Interventions: Other: Treatment as Usual (TAU) Only

INTERVENTIONS:
Behavioral: Internet-Based Cognitive Behavioral Therapy (ICBT) — An 8-week Internet-based Cognitive Behavioral Therapy (ICBT) program delivered via the National Health Research Institutes (NHRI) secure online platform. The program consists of 12 sequential modules released every 5 days, covering core CBT techniques such as cognitive restructuring, emotion regulation, behavioral activation, mindfulness, and self-compassion. Participants receive automated email notifications for new modules and supplementary review materials. Progress is monitored through the platform, and participants complete standardized self-report assessments at baseline, mid-intervention (week 5), post-intervention (week 9), and 3-month follow-up.
  Other Names: Online CBT; Web-based CBT
  Arms: TAU + ICBT
Other: Treatment as Usual (TAU) Only — Routine clinical care provided by a psychiatrist, which may include pharmacological treatment, psychoeducation, and regular follow-up visits according to clinical judgment. No ICBT intervention is provided during the study period. Participants follow the same assessment schedule as the experimental group. After the 3-month follow-up, participants in this group may request access to the ICBT program.
  Other Names: Standard Psychiatric Care
  Arms: TAU Only

SUMMARY:
This study aims to evaluate the effectiveness of internet-based cognitive behavioral therapy (ICBT) combined with treatment as usual (TAU) for adults diagnosed with generalized anxiety disorder (GAD) or major depressive disorder (MDD) in Taiwan.

CBT is a proven treatment for anxiety and depression, but traditional face-to-face sessions require frequent clinic visits, which may be costly and time-consuming. ICBT delivers similar therapy content online, allowing participants to complete sessions at their own pace, reducing barriers such as travel and scheduling.

A total of 160 participants will be randomly assigned to receive either TAU alone or TAU plus an 8-week ICBT program delivered via a secure national research platform. The program includes 12 online modules covering cognitive restructuring, emotion regulation, and behavioral activation techniques. Participants will complete assessments before, during, and after the program, with follow-up at 3 months.

The results will help determine whether ICBT can improve symptoms, enhance treatment accessibility, and support the integration of digital mental health interventions into clinical practice in Taiwan.

DETAILED DESCRIPTION:
This randomized controlled trial will assess the efficacy and feasibility of a locally adapted internet-based cognitive behavioral therapy (ICBT) program for patients with generalized anxiety disorder (GAD) or major depressive disorder (MDD) in Taiwan. The trial will be conducted at the Department of Psychiatry, National Taiwan University Hospital Hsin-Chu Branch, in collaboration with the National Health Research Institutes (NHRI).

A total of 160 eligible participants (aged 20-65 years) diagnosed with GAD or MDD will be recruited and randomly assigned to either the experimental group (TAU + ICBT) or the control group (TAU only), with 80 participants in each diagnostic category. The ICBT program lasts for 8 weeks and consists of 12 online modules, each released every 5 days, incorporating techniques such as cognitive restructuring, mindfulness, self-compassion, and behavioral activation. The control group will receive TAU and will be offered access to the ICBT program after study completion.

Assessments will be conducted at baseline, mid-intervention (week 5), post-intervention (week 9), and 3-month follow-up, using standardized self-report measures including GAD-7, PHQ-9, DASS-21, ISI, and other psychological well-being and user experience scales.

Primary outcomes are symptom reduction in anxiety (GAD-7) and depression (PHQ-9). Secondary outcomes include changes in psychological distress, insomnia severity, self-compassion, intolerance of uncertainty, and user satisfaction. Data will be analyzed using between-group comparisons and hierarchical linear modeling to evaluate both immediate and sustained intervention effects.

The study is expected to provide empirical evidence for the integration of digital mental health interventions into clinical practice, improve treatment accessibility, and support policy and service innovation in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 65 years.
* Diagnosis of Generalized Anxiety Disorder (GAD) confirmed by a psychiatrist.
* Diagnosis of Major Depressive Disorder (MDD) confirmed by a psychiatrist, without acute suicidal risk (screened by PHQ-9 Item 9; score of 3 requires further clinical assessment to exclude active suicidal plan or recent self-harm).

Exclusion Criteria:

* For GAD ICBT participants

  * Current or past history of obsessive-compulsive disorder, panic disorder, bipolar disorder, eating disorder, schizophrenia, or substance abuse.
  * Severe depressive symptoms impairing daily functioning.
  * Current suicidal ideation.
  * Experiencing acute life stressors (e.g., domestic violence, ongoing treatment for serious physical illness).
  * Currently receiving psychological counseling or psychotherapy.
  * Other serious factors limiting participation (e.g., intellectual disability, significant cognitive impairment, severe vision or hearing impairment).
* For MDD ICBT participants

  * Diagnosis of bipolar disorder, eating disorder, schizophrenia, psychotic symptoms, or substance abuse.
  * Current suicidal ideation or recent self-harm (PHQ-9 Item 9 score of 3 triggers further assessment; exclusion if active suicidal plan or recent self-harm present).
  * Experiencing acute life stressors (e.g., domestic violence, ongoing treatment for serious physical illness).
  * Currently receiving psychological counseling or psychotherapy.
  * Other serious factors limiting participation (e.g., intellectual disability, significant cognitive impairment, severe vision or hearing impairment).

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Generalized Anxiety Disorder symptoms (GAD-7 score) between intervention and control groups | Baseline, Week 5 (mid-intervention), Week 9 (post-intervention), and 3-month follow-up.
  The Generalized Anxiety Disorder-7 (GAD-7) is a 7-item self-report questionnaire assessing the severity of generalized anxiety symptoms over the past two weeks. Each item is scored from 0 ("not at all") to 3 ("nearly every day"), for a total score range of 0-21; higher scores indicate greater anxiety severity. The primary analysis will compare score changes from baseline to each follow-up point between the ICBT + Treatment as Usual (TAU) group and the TAU-only group.
Change in depressive symptoms (PHQ-9 score) between intervention and control groups | Baseline, Week 5 (mid-intervention), Week 9 (post-intervention), and 3-month follow-up.
  The Patient Health Questionnaire-9 (PHQ-9) is a 9-item self-report questionnaire assessing the severity of depressive symptoms over the past two weeks. Each item is scored from 0 ("not at all") to 3 ("nearly every day"), for a total score range of 0-27; higher scores indicate greater depression severity. The primary analysis will compare score changes from baseline to each follow-up point between the ICBT + TAU group and the TAU-only group.

OTHER OUTCOMES:
Course completion rate | Week 9 (post-intervention)
  The percentage of participants who complete all 12 modules of the Internet-based Cognitive Behavioral Therapy (ICBT) program within the 8-week intervention period. Completion is defined as accessing and finishing all module activities.
Platform usage metrics | Week 9 (post-intervention)
  Total number of logins and cumulative time spent on the ICBT platform during the intervention period, as recorded by the system's usage tracking function.
Changes in perception of online psychological interventions (POPII score) | Baseline, Week 9 (post-intervention), and 3-month follow-up
  The Perception of Online Psychological Intervention Index (POPII) is a self-developed questionnaire assessing perceived emotional support, knowledge and skill acquisition, self-awareness, and self-care practices after participation in ICBT. Higher scores indicate greater perceived benefit.